CLINICAL TRIAL: NCT05856981
Title: An Open-Label, Multicenter, Multi-arm Phase 1 Study Evaluating the Safety and Pharmacokinetics of ADU-1805 in Adults With Advanced Solid Tumors
Brief Title: Phase 1 Study Evaluating the Safety and PK of ADU-1805 in Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sairopa B.V. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SRP-22C102
Record Dates: First submitted 2023-01-04; First posted 2023-05-12 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-05

CONDITIONS: Solid Tumor, Adult; Metastatic Solid Tumor; Refractory Cancer; CRC, Colorectal Cancer; RCC, Clear Cell Adenocarcinoma; NSCLC (Advanced Non-small Cell Lung Cancer); Endometrial Cancer
Keywords: Immunotherapy
MeSH Terms: conditions — Neoplasm Metastasis; Neoplasms; Colorectal Neoplasms; Carcinoma, Renal Cell; Carcinoma, Non-Small-Cell Lung; Endometrial Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Monotherapy dose escalation, IV, Q3W, multiple dose levels (Experimental): ADU-1805 monotherapy dose escalation
  Interventions: Drug: ADU-1805
- Combination dose escalation, IV, Q3W, multiple dose levels, pembrolizumab at fixed dose (Experimental): ADU-1805 plus pembrolizumab dose escalation
  Interventions: Drug: ADU-1805; Drug: Pembrolizumab
- Combination dose expansion, IV, Q3W, multiple dose levels, pembrolizumab at fixed dose (Experimental): ADU-1805 plus pembrolizumab dose expansion
  Interventions: Drug: ADU-1805; Drug: Pembrolizumab

INTERVENTIONS:
Drug: ADU-1805 — anti-SIRPα monoclonal antibody
Drug: Pembrolizumab — Keytruda
  Other Names: Keytruda
  Arms: Combination dose escalation, IV, Q3W, multiple dose levels, pembrolizumab at fixed dose; Combination dose expansion, IV, Q3W, multiple dose levels, pembrolizumab at fixed dose

SUMMARY:
This first-in-human, open-label, multicenter, multi-arm dose-escalation study is designed to evaluate the safety, PK, and PD of ADU-1805, an anti- SIRPα monoclonal antibody, as monotherapy and in combination with pembrolizumab (anti-PD-1 antibody).

DETAILED DESCRIPTION:
This study is designed to evaluate the safety, PK, PD and preliminary clinical activity of ADU-1805, an anti- SIRPα monoclonal antibody, as monotherapy and in combination with pembrolizumab (anti-PD-1 antibody). The study is divided into a dose escalation phase and a dose expansion phase.

The dose expansion phase investigates ADU-1805 plus pembrolizumab at the respective recommended phase 2 dose (RP2D) in four advanced solid tumors: advanced PD-(L)1-naïve MSS colorectal cancer (CRC), PD-1 relapsed/refractory patients with either advanced MSS endometrial cancer (EC), renal cell carcinoma (RCC) or non-small cell lung cancer (NSCLC) patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged ≥18 years
* Signed and dated informed consent form
* Measurable disease according to RECIST (Safety Expansion only)
* ECOG Performance status of 0 or 1
* Adequate organ and marrow function
* Escalation Phase: Histologically and/or cytologically confirmed diagnosis of metastatic or unresectable solid tumors that are refractory to standard therapy or for which no standard therapy exists
* Expansion Phase: histologically and/or cytologically confirmed diagnosis of advanced PD-(L)1-naïve MSS colorectal cancer (CRC), PD-1 relapsed/refractory patients with either advanced MSS endometrial cancer (EC), renal cell carcinoma (RCC) or non-small cell lung cancer (NSCLC) patients, and that have measurable disease according to RECIST

Exclusion Criteria:

* Escalation Phase: Patients that suffer from melanoma, brain tumors, glioblastoma, sarcoma and pancreatic ductal adenocarcinoma (PDAC)
* Expansion Phase:

  * > 3 lines of prior systemic treatments
  * MSS colorectal cancer (CRC): liver metastasis present
* Pregnancy or breast-feeding
* Prior treatment with or receipt of:

  * biological agents, including monoclonal antibodies and immunotherapies, within 28 days prior to the first dose of ADU-1805
  * chemotherapy, targeted small molecule therapy, hormonal therapy or radiation therapy within 21 days prior to the first dose of ADU-1805 and within 42 days for nitrosoureas and mitomycin C.
  * anti-SIRPα or anti-CD47-directed therapy
  * systemic chronic steroid therapy or immunosuppressive therapy within 14 days prior to the first dose of ADU-1805
  * other investigational new drug or investigational device within 28 days prior to the first dose of ADU-1805
  * vaccine containing live virus within 28 prior to the first dose of ADU-1805
* Active untreated brain metastases
* Active infection requiring systemic therapy
* Impaired cardiac function or clinically significant cardiac disease
* Current Grade >2 toxicity related to prior anti-cancer therapy
* History of drug-induced severe immune-related adverse reaction
* Prior severe hypersensitivity to other monoclonal antibodies or ADU-1805 excipients
* Major surgery within defined period
* Diagnosis or positive test of HIV, hepatitis B, hepatitis C, or active tuberculosis
* Allogenic tissue/solid organ transplant
* Any intercurrent illness that is life-threatening or of such clinical significance that it would interfere with the patient's safety or ability to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2023-04-03 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Escalation Phase: Incidence and severity of dose limiting toxicity (DLT), treatment-emergent adverse events (TEAEs), and changes from baseline in safety parameters | First 21 days of treatment
  Incidence of DLTs and incidence and severity of TEAEs, classified according to NCI-CTCAE v. 5.0
Expansion Phase: Evaluate the clinical response of ADU-1805 plus pembrolizumab administered as an intravenous (IV) infusion. | Through study completion, up to 2,5 years
  Objective tumor response rate (ORR) per the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1

SECONDARY OUTCOMES:
Escalation and Expansion Phase: Pharmacokinetics of ADU-1805 monotherapy and ADU-1805 plus pembrolizumab, serum concentration-time profile and PK parameters | Through study completion, up to 2,5 years
  Serum concentration-time profiles and PK parameters (including Cmax, AUC)
Escalation and Expansion Phase: Immunogenicity of ADU-1805 monotherapy and ADU-1805 plus pembrolizumab | Through study completion, up to 2,5 years
  Incidence of anti-ADU-antibodies
Expansion Phase: To confirm safety of ADU-1805 in combination with pembrolizumab as an IV infusion | Through study completion, up to 2,5 years
  Incidence and severity of treatment-emergent adverse events (TEAEs), and changes from baseline in safety parameters.

OTHER OUTCOMES:
Escalation and Expansion Phase: Pharmacodynamics of ADU-1805 monotherapy and ADU-1805 plus pembrolizumab | Through end of treatment, up to 2 years
  Investigate the mechanism of action and pharmacodynamics (PD) of ADU-1805 monotherapy and ADU-1805 plus pembrolizumab using tumor tissue and blood biomarkers (e.g. immune monitoring)
Escalation and Expansion Phase: Preliminary Clinical activity of ADU-1805 monotherapy and ADU-1805 plus pembrolizumab | Through study completion, up to 2,5 years
  Overall and duration of response per (i)RECIST, PFS, (duration) of disease control, OS

CONTACTS AND LOCATIONS:
Locations (7):
- United States (4):
  - Henry Ford Cancer Institute, Detroit, Michigan
  - Washington University Medical Campus, St Louis, Missouri
  - Gabrail Cancer & Research Center, Canton, Ohio
  - Virginia Cancer Specialists, Fairfax, Virginia
- Grand Hopital de Charleroi (GHdC) - Hopital Notre Dame, Charleroi, Belgium
- Spain (2):
  - Hosp 12 de Octubre, Madrid
  - Hospital General Universitario Gergorio Maranon, Madrid

IPD SHARING:
Plan to Share IPD: No